CLINICAL TRIAL: NCT06377774
Title: To Optimize Therapeutic Procedures of Double-plasma Molecular Absorption System Therapy in acute-on Chronic Liver Failure Patients: a Prospective, Sigle Arm and Multicenter Study
Brief Title: To Optimize Therapeutic Procedures of DPMAS in ACLF Patients: a Prospective, Sigle Arm and Multicenter Study
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-096
Record Dates: First submitted 2024-04-14; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: double plasma molecular adsorption system; acute-on-chronic liver failure; short-term mortality
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The study will collect biological-samples including whole blood, urine and stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DPMAS therapy group: This is a prosepctive, sigle-arm and muticenter study. The study will enroll ACLF patients which receive the DPMAS therpay during hospitalization.
  Interventions: Other: No intervention in this study

INTERVENTIONS:
Other: No intervention in this study — No intervention in this study

SUMMARY:
Acute-on-chronic liver failure (ACLF) is a life-threaten syndrome carrying high-short-term mortality raging 40% to 60% within 90 days in patients with chronic liver disease. Double plasma molecular adsorption system (DPMAS) is one of the available artificial liver support systems, which combines plasma filtration and two specific adsorption membranes dedicating to remove bilirubin and the middle molecular toxins respectively. The efficiency of DMPAS treatment in liver failure patients remains controversial. Previous study indicate that liver failure patients with DPMAS therapy improve the short-term mortality and prevent the diseases progression within 28 days (PADSTONE Study). Thus, this single-arm, multicenter and prospective study is to further validate and optimize the therapeutic procedures of DPMAS therapy in ACLF patients.

DETAILED DESCRIPTION:
Liver failure in patients with chronic liver disease (CLD) and carries high short-term mortality ranging 40% to 60% within 90 days. In China Mainland, chronic hepatitis B virus (HBV) infection is the most common etiology of liver failure in CLD patients which reveals histological signature with submissive hepatic necrosis. While liver transplantation (LT) remains the treatment of choice, the lack of organ transplants necessitates finding alternative solutions. Supportive therapy including cardiovascular or renal support, treatment of encephalopathy and extracorporeal liver support, are the available treatments for liver failure patients in the clinical practice.

Artificial liver support system (ALSS) can remove inflammatory cytokines and toxins which is commonly used in clinical practice to treat liver failure. Double plasma molecular adsorption system (DPMAS) which is one of the ALSS combines plasma filtration and two specific adsorption membranes which can effectively remove bilirubin and the middle molecular toxins respectively. Within the last years, DPMAS is developed to one of the most recent non-biological extracorporeal liver support devices that used in acute or acute-on-chronic liver failure (ACLF) patients. In the clinical practice, DPMAS therapy in liver failure patients usually combines with therapeutic plasma exchange (PE). Previous investigations suggested that DPMAS and therapeutic PE were similar in improving 90-day survivals and DPMAS together with PE ameliorated the inflammatory response and improved the 28-day survival in HBV related ACLF.

However, the efficiency of DMPAS treatment in liver failure patients remains controversial and no large scale study to explore the potential subgroup of liver failure patients with chronic liver disease that may benefit from DPMAS therapy at present. Our previous study (PADSTONE Study) indicate that DPMAS therapy may improve the short-term mortality and prevent the disease progression in ACLF patients which needs to be further validated.

Accordingly, this single-arm study will enroll the ACLF patients with DPMAS therapy and aim to optimize and validate the therapeutic procedures of the DPMAS therapy in ACLF patients. Biological-samples will be collected in this study including plasma, urine and stools and multi-omics will be performed to explore and validate the precise profiles/biomarkers of the indication of DPMAS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent voluntarily;
2. Age>18 years old;
3. Inpatients;
4. Chronic liver disease;
5. The value of total bilirubin≥12mg/dl and INR≥1.5;
6. Patients are planned to have DPMAS therapy according to the physicians' judgment.

Exclusion Criteria:

1. The pregnant;
2. With severe chronic heart disease (NYHA>II);
3. With severe chronic obstructive pulmonary disease (GOLD>III);
4. With serious mental illness that prevents patients from sell-reporting;
5. Patients with unstable hemodynamics caused by infection or acute bleeding;
6. Diagnosis of hepatocellular carcinoma during screening period (BCLC>B);
7. With severe extrahepatic malignant carcinoma;
8. Patients who had liver resection or other organ transplantation;
9. Patients who had participated in, or are planning to participate in other clinical trial within the 3 months prior to enrollment;
10. Hospital stays <48 hours;
11. Not suitable to participate in this study judging by researchers;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focus on acute-on-chronic liver failure (ACLF) patients which carries high prevalence and short-term mortality. ACLF patients are featured by multiple organ failure. Except for liver transplantation, the routine use of artificial or bioartifical extracorporeal liver support or plasma exchange appears to be a promising and effective bridging therapy in patients with ACLF to liver transplantation or spontaneous regeneration.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
28-day transplantation-free mortality | 28 days
  Comparing to the PADSTONE study, the 28-day transplantation-free mortality in ACLF patients with DPMAS therapy.
The disease progression rate | 28 days
  Comparing to the PADSTONE study, the disease progression (progress to EASL defined ACLF) rate within 28 days.

SECONDARY OUTCOMES:
the 90-day transplantation-free mortality | 90 days
  Comparing to the PADSTONE study, the 90-day transplantation-free mortality in ACLF patients with DPMAS therapy.
the disease progression | 90 days
  Comparing to the PADSTONE study, the disease progression (progress to EASL defined ACLF) rate within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinjun Chen, Dr., Principal Investigator — Nanfang Hospital, Southern Medical University

IPD SHARING:
Plan to Share IPD: No